CLINICAL TRIAL: NCT01550731
Title: Preparing Older Veterans With Serious and Chronic Illness for Decision Making
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IIR 11-110
Record Dates: First submitted 2011-12-08; First posted 2012-03-12 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-05

CONDITIONS: Aging
Keywords: advance care planning; health communication; aging
MeSH Terms: interventions — Advance Directives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREPARE (Experimental): The intervention group will review the PREPARE advance care planning website and PREPARE materials plus receive an advance directive. The control group will only receive an advance directive.
  Interventions: Behavioral: PREPARE website
- CONTROL (Active Comparator): The control group will only receive an advance directive.
  Interventions: Behavioral: Advance directive

INTERVENTIONS:
Behavioral: PREPARE website — Advance care planning website and materials plus an advance directive.
  Arms: PREPARE
Behavioral: Advance directive — The control group will only receive an advance directive.
  Arms: CONTROL

SUMMARY:
Millions of diverse Veterans live with severe and chronic illness for which they will face complex, ongoing decisions. Although the VHA has been at the forefront of patient-centered chronic care, interventions to prepare Veterans for complex decision-making over the course of chronic illness are lacking. This proposal addresses this gap by testing the efficacy of a novel preparation guide designed to prepare Veterans to communicate with their surrogates and to work with clinicians to make complex, ongoing decisions. The multi-media guide teaches communication and preparation skill behaviors (e.g., how to choose a surrogate and ask clinicians questions) in a culturally appropriate, easy-to-use format (targeted to a 5th grade reading level). This study aims to provide an impetus for changing the paradigm of advance care planning policies within the VA by moving beyond documentation of end-of-life wishes to the activation of Veterans to participate in ongoing communication of their values and goals - a process that is essential to fully realize patient-centered care.

DETAILED DESCRIPTION:
4.5 million Veterans are over age 65 and an increasing number are living with chronic and serious illness. Most older Veterans and their surrogate decision makers will eventually face complex, ongoing decisions over the course of chronic illness. These decisions are difficult, especially for the 50% of older Veterans with limited health literacy. The old paradigm of advance care planning has focused on making decisions about life- prolonging procedures (e.g., resuscitation) by completing advance directives. Yet, this old paradigm is problematic. The forms are difficult to understand and often culturally insensitive. They also fail to prepare patients with concrete skills, such as how to identify one's values and communicate with surrogates and clinicians. The investigators have published a new paradigm of advance care planning that focuses instead on preparing patients to communicate with their surrogates and to actively participate with clinicians in making the best possible in-the-moment decisions. The new paradigm seeks to ensure that complex, ongoing decisions are based on a comprehensive set of considerations including the current clinical context, evolving goals, and patients' and surrogates' needs. To do this effectively, Veterans need to prepare. However, an easy-to-use, culturally-appropriate preparation guide does not exist. The investigators have created an easy-to-understand (5th grade reading level) preparation guide based on the investigators' new paradigm called PREParation, Activation, Reflection, and Engagement in advance care planning or PREPARE. PREPARE is designed to teach Veterans preparation skills including how to choose a surrogate and discuss surrogate decision making, clarify personal values for specific health states, and ask clinicians questions to make informed choices. The aims of this study are: (1) to conduct a randomized control trial to determine the efficacy of PREPARE to engage older Veterans with chronic illness in preparation skill behaviors (i.e., did they choose a surrogate, clarify their values, ask clinicians questions); (2) to determine the efficacy of PREPARE to activate Veterans and clinicians within clinical encounters (i.e., did Veterans ask clinicians questions or discuss preparation topics and did clinicians respond) and to improve satisfaction with decision making; and (3) to obtain input from Veterans, surrogates, and clinicians about implementation of PREPARE within the VA. To achieve Aim 1, 205 Veterans will be randomly assigned to the intervention (PREPARE materials plus an advance directive) and 205 will be assigned to the control group (advance directive only). Veterans in the PREPARE arm will view the easy-to-understand, multi-media PREPARE website during the study interview and then take home PREPARE materials in photo booklet and pamphlet format to ensure universal access to the information. The primary outcome is Veteran-reported engagement in preparation skill behaviors at 3 and 6 months, which will be measured with standard cognitive behavioral measures. For Aim 2, activation within the clinical encounters will be measured with validated quantitative analysis techniques of audio-recordings. Satisfaction with decision making will be measured with validated, self-reported measures. For Aim 3, the investigators will ask Veterans randomized to the PREPARE arm and their surrogates and clinicians how best to implement PREPARE within the clinical setting. The investigators will use standard parametric or non-parametric statistical tests to assess group differences, will control for demographic or other variables that differ between randomization groups, and adjust for potential clustering by clinician. For Aims 1 and 2 the investigators will assess differences in engagement and satisfaction by race/ethnicity, literacy, and gender. The research team has extensive experience testing literacy-appropriate, multi-media health education materials in randomized trials. The study team is poised to test the efficacy of PREPARE, and findings from this study will pave the way for multi-site effectiveness testing and widespread VA dissemination of PREPARE.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* 60 years of age
* who have been seen in the General Medicine, Geriatrics, and Women's Clinics twice in the past year
* and have 2 or more serious or chronic medical conditions as determined by ICD-9 codes

Exclusion Criteria:

* Veterans will be excluded if they are:

  * deaf
  * blind
  * demented

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2012-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sudore, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McMahan RD, Knight SJ, Fried TR, Sudore RL. Advance care planning beyond advance directives: perspectives from patients and surrogates. J Pain Symptom Manage. 2013 Sep;46(3):355-65. doi: 10.1016/j.jpainsymman.2012.09.006. Epub 2012 Nov 27. PMID 23200188
- [Result] Allison TA, Sudore RL. Disregard of patients' preferences is a medical error: comment on "Failure to engage hospitalized elderly patients and their families in advance care planning". JAMA Intern Med. 2013 May 13;173(9):787. doi: 10.1001/jamainternmed.2013.203. No abstract available. PMID 23545699
- [Result] Sudore RL, Knight SJ, McMahan RD, Feuz M, Farrell D, Miao Y, Barnes DE. A novel website to prepare diverse older adults for decision making and advance care planning: a pilot study. J Pain Symptom Manage. 2014 Apr;47(4):674-86. doi: 10.1016/j.jpainsymman.2013.05.023. Epub 2013 Aug 21. PMID 23972574
- [Result] Sudore RL, Stewart AL, Knight SJ, McMahan RD, Feuz M, Miao Y, Barnes DE. Development and validation of a questionnaire to detect behavior change in multiple advance care planning behaviors. PLoS One. 2013 Sep 5;8(9):e72465. doi: 10.1371/journal.pone.0072465. eCollection 2013. PMID 24039772
- [Result] Su CT, McMahan RD, Williams BA, Sharma RK, Sudore RL. Family matters: effects of birth order, culture, and family dynamics on surrogate decision-making. J Am Geriatr Soc. 2014 Jan;62(1):175-82. doi: 10.1111/jgs.12610. Epub 2014 Jan 2. PMID 24383459
- [Result] Sudore R, Le GM, McMahan R, Feuz M, Katen M, Barnes DE. The advance care planning PREPARE study among older Veterans with serious and chronic illness: study protocol for a randomized controlled trial. Trials. 2015 Dec 12;16:570. doi: 10.1186/s13063-015-1055-9. PMID 26654250
- [Result] Sudore RL, Boscardin J, Feuz MA, McMahan RD, Katen MT, Barnes DE. Effect of the PREPARE Website vs an Easy-to-Read Advance Directive on Advance Care Planning Documentation and Engagement Among Veterans: A Randomized Clinical Trial. JAMA Intern Med. 2017 Aug 1;177(8):1102-1109. doi: 10.1001/jamainternmed.2017.1607. PMID 28520838
- [Derived] Lum HD, Barnes DE, Katen MT, Shi Y, Boscardin J, Sudore RL. Improving a Full Range of Advance Care Planning Behavior Change and Action Domains: The PREPARE Randomized Trial. J Pain Symptom Manage. 2018 Oct;56(4):575-581.e7. doi: 10.1016/j.jpainsymman.2018.06.007. Epub 2018 Jun 27. PMID 29940209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans were enrolled from a women's, geriatrics, and several general medicine clinics at the San Francisco VA from April 2013 through July 2016. Veterans had to be 60 years or older, have had at least 2 chronic medical conditions, and had 2 or more visits with a primary care clinician, plus 2 VA clinic, ER, or hospital visits in the past year.
Period: Overall Study
Arm/Group | PREPARE | CONTROL
Started | 205 | 209
Completed | 205 | 209
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREPARE | CONTROL | Total
Number analyzed (Participants) | 205 | 209 | 414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 50 | 96
  >=65 years | 159 | 159 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (7.7) | 71.5 (7.9) | 71.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 186 | 190 | 376
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 33
  Not Hispanic or Latino | 189 | 192 | 381
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 46 | 42 | 88
  White | 129 | 139 | 268
  More than one race | 14 | 12 | 26
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 205 | 209 | 414

OUTCOME MEASURES:

1. Primary Outcome: New Advance Care Planning Documentation in the Medical Record at 9 Months
Description: The primary outcome is documentation of advance care planning wishes in the medical record. ACP documentation for the purposes of this study includes the easy-to-read advance directive or other valid advance directives or living wills, a durable power of attorney for healthcare document (DPOAHC), a physicians orders for life sustaining treatment (POLST) form, or other documentation of patients wishes for medical care (ie, documentation of oral directives by a physician, or code status, such as full code or do not resuscitate or do not intubate orders or notes by a physician).
Time Frame: 9 months after study enrollment
Measure: Number; unit: percentage of participants
Arm/Group | PREPARE | CONTROL
Number analyzed (Participants) | 205 | 209
percentage of participants | 35 | 25

2. Secondary Outcome: Self-reported Engagement in Advance Care Planning (ACP) Behaviors
Description: Secondary outcome was chosen to measure the full process of Advance Care Planning (ACP) using validated questionnaires, such as the patient-reported ACP Engagement Survey. This questionnaire includes Behavior Change Process measures. Behavior Change Process measures include knowledge, contemplation, self-efficacy, and readiness for several ACP actions. The Process measures are assessed on an average 5-point Likert scale with a low of 1 and a high of 5, with high scores indicating more ACP engagement. The investigators used mixed effects models to create an overall adjusted score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PREPARE | CONTROL
Number analyzed (Participants) | 205 | 209
score on a scale | 3.78 (3.67) | 3.64 (3.53)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the length of the study for each participant (6 months).
Description: For this behavioral trial, adverse events were defined as any unexpected negative psychological effects caused by the patient education materials.
Arm/Group | PREPARE | CONTROL
All-Cause Mortality (participants affected / at risk) | 0/205 | 0/209
Serious Adverse Events (participants affected / at risk) | 0/205 | 0/209
Other Adverse Events (participants affected / at risk) | 0/205 | 0/209

LIMITATIONS AND CAVEATS:
Older veterans were recruited from clinics at the SFVA, potentially limiting generalizability. Materials were viewed in study offices with computer access, potentially limiting generalizability. Study interviews and reminder calls may be activating.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes